CLINICAL TRIAL: NCT01624376
Title: A Randomized, Double-blind, Placebo-controlled Phase I/IIa Study in Patients With Abdominal or Perianal Fistulizing Crohn's Disease to Explore the Safety, Tolerability and Preliminary Efficacy of Locally Administered DLX105.
Brief Title: Randomized, Double-blind, Placebo-controlled Study in Patients With Fistulizing Crohn's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Delenex Therapeutics AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DLX105-004-001-001
Record Dates: First submitted 2012-06-14; First posted 2012-06-20 (Estimated); Last update posted 2014-02-04 (Estimated); Status verified 2014-02

CONDITIONS: Fistulizing Crohn's Disease
Keywords: non-invasive management; Fistula; Crohn's Disease; local administration; non-invasive
MeSH Terms: conditions — Fistula; Crohn Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- DLX105 (Active Comparator): DLX105 local injection into the identified fistula(s)
  Interventions: Drug: DLX105
- Placebo Injection (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DLX105 — 10mg DLX105/injection injected into the fistula over a treatment period of 4 weeks.
  Arms: DLX105
Drug: Placebo — Placebo injections are administered over the treatment period of 4 weeks.
  Arms: Placebo Injection

SUMMARY:
The primary objective of this study is to investigate the safety and tolerability of locally administered DLX105 in treating enterocutaneous fistulas in Crohn's Disease patients.

The study will consist of a screening period of approx. 2 weeks, a 4-week treatment period and a 2-week follow-up period. An end-of study visit is scheduled on Day 43, 2 weeks after the last study visit.

DETAILED DESCRIPTION:
Beside investigation of the safety and tolerability of locally administered DLX105, the purpose of the study is also to evaluate the response rate and time to response of enterocutaneous fistulas following local injection of DLX105 (secondary objective).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Crohn' Disease
* Single or multiple enterocutaneous abdominal and/or perianal and/or rectovaginal fistulas of at least 3 months'duration.
* TNF-blocker naive patients or patients who are primary or secondary anti-TNF non-responders

Exclusion Criteria:

* CDAI greater than 450
* ongoing treatment with TNF-blockers (duration of wash-out prior to randomization is 8 weeks)
* Active abscess formation within fistula
* Abdominal or anorectal surgery within the last 4 weeks prior to randomization
* Known immunosuppression
* Infections, sepsis
* Positive Test for hepatitis B or C and HIV
* Patients who had life vaccination within 6 weeks prior first study drug administration, or will require live vaccination during the course of the trial
* Active liver disease with ALT and/or AST greater than 3x upper limit of normal
* Any severe, progressive or uncontrolled medical condition that in judgment of investigator prevents the patient from participating in the study.
* History or evidence of drug or alcohol abuse within the 6 months prior first study drug administration
* Pregnant or nursing women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive B-hCG laboratory test

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-06; Primary Completion 2013-02 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Local Tolerability | each study visit after randomization over a period of 4 weeks
  Investigator and Patient will assess the local tolerability of DLX105 for each treated fistula using a 10-cm visual analogue scale (VAS) at each study visit. Changes from Baseline will be reported descriptively.
Reduction of Number of draining fistulas | Day 29 and Day 43 after randomization
  Reduction of number of draining fistulas of 50% from baseline observed at Visit 10 and confirmed at End of Study Visit.

SECONDARY OUTCOMES:
Complete Response | Day 29 and Day 43 after randomization
  Complete absence of drainage from all of the fistulas treated in a given patient despite gentle finger compression
Perianal Disease Activity Index (PDAI) Score | Baseline, Day 15, Day 29, Day 43 after randomization
  Evaluate the efficacy with completion of PDAI at the given visits.
Number of Participants with Adverse Events as a Measure of Safety and Tolerapility | each study visit over a period of 6 weeks after randomization

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Zurich, Switzerland